CLINICAL TRIAL: NCT06975514
Title: A Randomized, Double-blind, Active-controlled, Parallel-group Clinical Study to Evaluate the Efficacy and Safety of YZJ-1139 Tablets in the Treatment of Insomnia Disorder
Brief Title: Safety and Efficacy Study of YZJ-1139 Tablets in Insomnia Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YZJ-1139-3-02
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YZJ-1139 group (Experimental)
  Interventions: Drug: YZJ-1139
- Zolpidem group (Active Comparator)
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: YZJ-1139 — YZJ-1139 20mg tablets, once daily in the evening
  Arms: YZJ-1139 group
Drug: Zolpidem — Zolpidem 10mg tablets, once daily in the evening
  Arms: Zolpidem group

SUMMARY:
The main purpose of this study is to assess efficacy of YZJ-1139 for 28 days in adult subjects with insomnia disorder. Efficacy will be evaluated on objective and subjective sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, aged ≥ 18 to < 65 years.
2. Meet the clinical diagnostic criteria for insomnia disorder as defined in ICSD-3 criteria.
3. sTSO ≥ 30 min for at least 3 nights per week and/or sWASO ≥ 60 min for at least 3 nights per week within 4 weeks prior to screening.
4. Able to recognize 26 English letters and MMSE score indicats no cognitive impairment.
5. During the run-in period and on Day 1 of the treatment period, sTSO ≥ 30 min for at least 3 nights in the last 7 sleep diaries and/or sWASO ≥ 60 min for at least 3 nights out of 7 nights as confirmed by the sleep diary prior to PSG monitoring.
6. PSG results for 2 consecutive nights during the run-in period should meet the following conditions:

   1. The mean LPS ≥ 30 min for 2 nights and ≥ 20 min for any one night; And/or the mean WASO ≥ 60 min for 2 nights, and ≥ 45 min either night.
   2. The mean SE ≤ 85% for 2nights, with the SE ≤ 87.5% for both nights .
7. ISI score ≥ 15 at screening and on Day 1 of the treatment period .
8. Have a bedtime between 9 p.m. and 1 a.m., wake up between 5 a.m. and 10 a.m., and stay in bed for 6.5 to 9 hours for at least 5 nights in the last 7 sleep diaries as confirmed by the sleep diary prior to PSG monitoring during the run-in period and on Day 1 of the treatment period.
9. Reproductive-age male and female participants must agree to use effective contraceptive measures from the screening visit through at least 30 days after the last dose of double-blind study treatment, and must not be planning to become pregnant or donate sperm/eggs during this period.
10. Understand the study procedures and contents, voluntarily participate in the clinical study and sign the written Informed Consent Form, have good compliance during participation in the study, and are willing to attend the visits.

Exclusion Criteria:

1. Hypersensitivity to YZJ-1139 tablets or zolpidem or to their excipients.
2. Have serious endocrine diseases, hematological diseases, cardiovascular and cerebrovascular diseases, gastrointestinal diseases, liver and kidney diseases, autoimmune diseases, impaired respiratory function or other related diseases, or have other medical history that may affect the safety of the subjects or interfere with the study assessments in the opinion of the investigator.
3. Have insomnia disorder due to other causes such as chronic pain, headache, eczema, neurodermatitis, allergic rhinitis, and serious dermatitis (difficulty sleeping due to physical reasons, difficulty falling asleep due to medical reasons).
4. Current or previous history of psychiatric or neurological disease such as epilepsy, schizophrenia, bipolar mental disorder, neurodevelopmental retardation, and cognitive disorder, or previous history of other mental illness that may affect the safety of the subjects or interfere with the study assessments in the opinion of the investigator.
5. Previous history of sleep-related respiratory disorders including obstructive sleep apnea (with or without continuous positive airway pressure [CPAP] therapy), periodic limb movement disorder, myasthenia gravis, restless legs syndrome, circadian rhythm sleep disturbances, narcolepsy or other sleep disorders: subjects with restless legs syndrome which is diagnosed by relevant diagnostic and treatment guidelines should be excluded. Those who have been cured of the above diseases can be enrolled.
6. Have previous complex sleep behaviors, such as sleep driving, sleep eating, and sleep phone calls.
7. Have nocturia increased caused by urinary tract infection, urinary tract injury or prostatic disorder.
8. Hyperthyroidism.
9. History of alcohol abuse (defined as regular daily alcohol consumption exceeding the following criteria: approximately 720 mL of beer, or 240 mL of wine, or 60 mL of liquor) within the past 6 months.
10. Regular daily consumption of excessive tea and coffee drinks (defined as consumption of > 4 cups of caffeinated beverages or > 400 mg of caffeine per day), or daily habituation to drinking caffeinated beverages beyond 18:00.
11. Exclusion Criteria: Smokers who have smoked more than 10 cigarettes per day within 6 months prior to screening or smokers who are unable to refrain from falling asleep.
12. Have any lifestyle that interferes with the study process or may interfere with sleep: for example, there will be travels across 3 or more time zones (mainland China is considered as 1 time zone) within the next 2 weeks or during the study period, or there will be shift work (night and daytime shift).
13. History of drug abuse within the past 2 years, or positive urine drug screening for any indicator; history of drug taking or addiction, which is known through questioning.
14. Have received any hypnotics, antidepressants, antipsychotic drugs, anticholinergics, memory-enhancing drugs, antihistamines, centrally acting analgesics, centrally acting muscle relaxants, central nervous system stimulants, CYP3A inducers, CYP3A inhibitors, traditional Chinese medicines and traditional Chinese medicinal products with sleep-improving effects, or any other therapies for insomnia disorder within 1 week prior to the run-in period or within 5 half-lives of the investigational product, whichever is longer.
15. Plan to undergo surgery during the study.
16. Depression: Hamilton Depression Scale (HAMD) score ≥ 18; anxiety: Hamilton Anxiety Scale (HAMA) score ≥ 14.
17. Suicidal ideation with or without plan at screening or within 6 months prior to screening (score ≥ 3 on item 3 [suicide] of HAMD, or select "Yes" on item 3, 4 or 5 of suicidal ideation subscale of C-SSRS), or have any suicidal behavior in the past 10 years (as assessed by the suicidal ideation subscale of C-SSRS).
18. ECG at screening shows QTcF interval prolongation (QTcF > 450 ms, QTcF=QT/(RR^0.33)).
19. AST or ALT > 2 × the upper limit of normal (ULN), or Cr > 1.5 × ULN.
20. Known to be human immunodeficiency virus (HIV) antibody positive at screening.
21. Apnea-hypopnea index [AHI] or periodic limb movement index [PLMI] > 10 times/hour detected by PSG monitoring during the run-in period.
22. Unable to avoid vaccination within 1 month prior to screening.
23. Enrolled in another clinical trial and used any investigational drug within 1 month or 5 half-lives (whichever is longer) prior to the run-in period, or participation in another investigational trial at the same time during this trial.
24. Previously participated in any clinical trial of YZJ-1139; or treated with other orexin receptor antagonists of appropriate amount and sufficient duration and who, in the opinion of the investigator, have failed treatment due to efficacy or safety.
25. Pregnant or lactating women.
26. Have other conditions that make the subject unsuitable for participation in the clinical study in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Mean Objective Wake After Sleep Onset (WASO) | Baseline, Day 1/Day 2, Day 27/Day 28
  WASO is defined as minutes of wake from the onset of persistent sleep until lights on as measured by polysomnography (PSG).
Change from baseline of Mean Objective Sleep Efficiency (SE) | Baseline, Day 1/Day 2, Day 27/Day 28
  SE is defined as percentage of time spent in bed asleep, calculated as total sleep time (TST) divided by interval from lights off until lights on as measured by PSG, multiplied by 100.
Change from baseline of Mean Objective Total Sleep Time (TST) | Baseline, Day 1/Day 2, Day 27/Day 28
  TST is defined as total sleep time measured by PSG.
Change from baseline of Mean Objective Latency to Persistent Sleep (LPS) | Baseline, Day 1/Day 2, Day 27/Day 28
  LPS is defined as latency to persistent sleep measured by PSG.

SECONDARY OUTCOMES:
Change from baseline of Mean Subject Wake After Sleep Onset (sWASO) | Baseline, Week1, Week 4
  sWASO is self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Change from baseline of Mean Subject Sleep Efficiency (sSE) | Baseline, Week1, Week 4
  sSE is defined as percentage of time spent in bed asleep, calculated as subject total sleep time (sTST) divided by interval from lights off until lights on, multiplied by 100.
Change from baseline of Mean subject Total Sleep Time (sTST) | Baseline, Week1, Week 4
  sTST is self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Change from baseline of Mean Subjective Time to Sleep Onset (sTSO) | Baseline, Week1, Week 4
  sTSO is self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Change from baseline of Mean Subjective Number of awakenings (sNAW) | Baseline, Week1, Week 4
  sNAW is self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Change from baseline of Sleep structure (wakefulness, N1, N2, N3, rapid eye movement sleep [REM], non-rapid eye movement sleep [NREM]) | Baseline, Day 1/Day 2, Day 27/Day 28
  Wakefulness, N1, N2, N3, REM, NREM are measured by PSG in minutes, and expressed as the percent change from time spent in bed (TIB) and TST.
Change from baseline of Sleep structure (REM latency, number of awakenings [NAW], arousal index for REM and NREM) | Baseline, Day 1/Day 2, Day 27/Day 28
  REM latency, NAW and the arousal index for REM and NREM are measured by PSG.
Change from baseline in the mean subjective sleep quality score | Baseline, Week1, Week 4
  Subjective sleep quality score is a self-report assessment of participant perception of the effects of a medication on their sleep. Higher score indicated severe insomnia problem.
Change from baseline in the ISI score | Baseline, Day15 and Day 28
  Insomnia Severity Index is a self-report questionnaire assessing the nature, severity, and impact of insomnia. Higher score indicated severe insomnia problem.
Percentage of participants on each scale of Global Impression of Insomnia (PGI-I) each item | Day15 and Day 28
  the PGI-I was a self-report assessment of participant perception of the effects of a medication on their sleep. The PGI-I had 3 items related to study medication effects (a) helped/worsened sleep, (b) decreased/increased time to fall asleep, (c) increased/decreased total sleep time, and 1 item related to perceived appropriateness of study medication strength. The first 3 items were answered on a 3-point scale (1=positive medication effect, 2=neutral medication effect, 3=negative medication effect) and the last item on a different 3 point scale (medication: 1=too strong, 2=just right, 3=too weak).

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Peking University People's Hospital, Beijing
  - ChengDu Second People's Hospital, Chengdu
  - ChongQing Traditional Chinese Medicine Hospital, Chongqing
  - Deyang People's Hospital, Deyang
  - The First Affiliated Hospital of Jinan University (Guangzhou Overseas Chinese Hospital), Guangzhou
  - The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital), Jinan
  - The Second Affiliated Hospital Of NanChang University, Nanchang
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - ShengJing Hospital Of China Medical University, Shenyang
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - SuZhou GuangJi Hospital, Suzhou
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Anding Hospital, Tianjin
  - Wuhan No.1 Hospital, Wuhan
  - Yan'an University Xianyang Hospital, Yan’an
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou